CLINICAL TRIAL: NCT01324466
Title: A Randomized, Double-Blind, Parallel-Group, Vehicle-Controlled, Multicenter Study of NB-001 in the Treatment of Recurrent Herpes Labialis
Brief Title: A Multicenter Study of NB-001 in the Treatment of Recurrent Herpes Labialis (SHaRCS)
Acronym: SHaRCS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NanoBio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NB-001-005
Record Dates: First submitted 2011-03-22; First posted 2011-03-29 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Recurrent Herpes Labialis
MeSH Terms: conditions — Herpes Labialis | interventions — 5-((2-(6-Amino-9H-purin-9-yl) ethyl) amino)-1-pentanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vehicle (Placebo Comparator): Vehicle
  Interventions: Drug: Vehicle
- Active (Active Comparator): Active NB-001(0.3%)
  Interventions: Drug: NB-001

INTERVENTIONS:
Drug: NB-001 — Topical, 5 times daily until investigator assessment of healing or a maximum of 4 days
  Arms: Active
Drug: Vehicle — Topical, 5 times daily until investigator assessment of healing or a maximum of 4 days
  Arms: Vehicle

SUMMARY:
The purpose of this study is to demonstrate the safety and efficacy of NB-001 in subjects with recurrent herpes labialis (RHL).

DETAILED DESCRIPTION:
This is a randomized, double-blind, two arm, parallel-group, vehicle-controlled, multi-center study of NB-001. The study is designed to demonstrate the safety and efficacy of NB-001 in subjects with RHL. Approximately 850 subjects who meet all eligibility criteria will be randomized in the study. Subjects will begin treatment as soon as they experience the onset of cold sore symptoms. Treatment will be applied 5 times daily, approximately 3-4 hours apart while awake. Treatment will continue until the investigator assesses the primary lesion complex as healed or a maximum of 4 days.

Clinic visits will occur on a daily basis until the investigator determines that the primary lesion complex has healed or a maximum of 15 clinic visits. At daily clinic visits, the investigator will make efficacy assessments of the primary lesion complex; safety and tolerability assessments of NB-001 following topical administration will also be assessed daily. Subjects will make daily assessments of therapy.

At the End of Study, the investigator will make a global assessment of therapy. The subject will make global assessments of therapy and social impact.

ELIGIBILITY:
Inclusion Criteria:

* A healthy man or woman 18 years of age or older. Women who are pregnant, lactating or may become pregnant may (at the investigator's discretion) be included in the study.
* Have recurrent herpes labialis as defined by a history of three (3) or more cold sore recurrences on the lips and/or skin surrounding the lips in the previous 12 months;
* Have the majority of their cold sore recurrences preceded by a well defined history of prodromal symptoms.

Exclusion Criteria:

* Subjects with severe chronic illness
* Received (within the last 6 months) or receiving chemotherapy;
* Significant skin disease on the face
* Previously received herpes vaccine;
* Active alcohol or drug abuse;
* Prior randomization into any NanoBio study;
* Known allergies to topical creams, ointments or other topical medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 847 (Actual)
Dates: Start 2011-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Time of Healing of the primary lesion complex | Median time to healing (day 1 until up to 4 days)
  Time to healing of the primary lesion complex (in days or fraction thereof) as assessed by the investigator. Time to healing is the time from application of the first dose to investigator assessed healing

SECONDARY OUTCOMES:
Proportion of subjects in whom the primary lesion complex does not progress beyond the Papule/Edema Stage. | First Post-Treatment Visit (after maximum 15 clinical visits)
  Proportion of subjects in whom the primary lesion complex does not progress beyond the Papule/Edema Stage. This analysis will be performed in the cohort of subjects whose primary lesion complex is assessed as being in the Prodrome (pain, burning, tingling, itching, redness, swelling, or a tight sensation of the lip), Erythema/Macule, Papule/Edema, or Aborted Stage by the investigator at the first post-treatment visit.

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Radiant Research, Inc., Birmingham, Alabama
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Radiant Research, Inc, Tucson, Arizona
  - Providence Clinical Research, Burbank, California
  - Axis Clinical Trials, Los Angeles, California
  - Staywell Research, Northridge, California
  - Front Range Clinical Research, Wheat Ridge, Colorado
  - Tampa Bay Medical Research, Clearwater, Florida
  - Altus Research, Inc., Lake Worth, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Radiant Research, Inc, Pinellas Park, Florida
  - Radiant Research, Inc. Chicago, Chicago, Illinois
  - DermResearch, Louisville, Kentucky
  - Commonwealth Biomedical Research, Madisonville, Kentucky
  - The Center for Pharmaceutical Research, P.C., Kansas City, Missouri
  - Radiant Research, Inc., St Louis, Missouri
  - Meridian Clinical Research, Omaha, Nebraska
  - Axis Clinical Trials, New Hyde Park, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - Radiant Research, Inc., Akron, Ohio
  - Radiant Research, Inc., Cincinnati, Ohio
  - Paramount Clinical Research, Bridgeville, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Radiant Research, Inc., Anderson, South Carolina
  - DermResearch, Inc., Austin, Texas
  - Research Across America, Dallas, Texas
  - Benchmark Research - San Angelo, San Angelo, Texas
  - Radiant Research, Inc., San Antonio, Texas
  - Utah Clinical Trials, LLC, Salt Lake City, Utah
  - South Valley Dermatology, West Jordan, Utah
  - IntegraTrials, LLC, Arlington, Virginia
  - National Clinical Research, Richmond, Virginia
  - Dermatology & Laser Center NW, Bellingham, Washington